CLINICAL TRIAL: NCT01970644
Title: Neurocognition After Gamma Knife Radiosurgery for Multiple Brian Metastases
Status: Terminated | Type: Observational
Why Stopped: Poor accrual. Investigator decision.
Sponsor: CancerCare Manitoba (Other)
Collaborators: Health Sciences Centre Foundation, Manitoba (Other)
Responsible Party: Sponsor
Other Study IDs: B2013:129
Record Dates: First submitted 2013-10-23; First posted 2013-10-28 (Estimated); Last update posted 2016-05-30 (Estimated); Status verified 2016-05

CONDITIONS: Neoplasm Metastases
Keywords: Neoplasm metastasis; Brain neoplasms; Radiosurgery; Cognition disorders; Cranial irradiation
MeSH Terms: conditions — Neoplasm Metastasis; Brain Neoplasms; Cognition Disorders | interventions — Radiosurgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Brain metastases (>= 4): Patients with pathologically proven solid tumour malignancy who have >=4 brain metastases will be treated with gamma knife radiosurgery.
  Interventions: Radiation: Gamma knife radiosurgery

INTERVENTIONS:
Radiation: Gamma knife radiosurgery — Depending on maximum tumour diameter, patients will receive a single dose of 15-20 Gy to the isodose surface which encompasses the entire metastasis.

SUMMARY:
Cancer which spreads to the brain (brain metastases) is a common and significant problem. Historically, whole-brain radiotherapy has been used to treat these patients but has a negative effect on cognition. Radiosurgery is an alternative treatment with potential for fewer cognitive side effects. The impact of radiosurgery alone on the cognitive function of patients with multiple brain metastases is not well studied. We propose a pilot study at the Winnipeg Centre for Gamma Knife Surgery to examine this issue.

DETAILED DESCRIPTION:
Patients with >=4 brain metastases will undergo Gamma Knife radiosurgery to a dose of 15-20 Gy, depending on the maximum tumour diameter and number of metastases. A number of neurocognitive, quality of life, and toxicity assessments will be performed at baseline and at 6 weeks post-radiosurgery, then at months 4, 6, 12, 18, and every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically proven solid tumour malignancy
* Age >= 18 years
* Karnofsky performance status >= 70
* >= 4 brain metastases, all eligible to be treated with radiosurgery
* All brain metastases <= 4.0 cm in any diameter
* Pre-treatment contrast enhanced MRI brain <= 42 days prior to enrollment
* Patient able to provide his/her own written informed consent

Exclusion Criteria:

* Prior radiosurgery, whole brain radiotherapy, or cranial radiotherapy
* Previous surgical resection of brain metastasis (biopsy is allowed)
* Prior chemotherapy ≤ 7 days prior to enrollment
* Planned chemotherapy during radiosurgery
* Leukemia, lymphoma, germ-cell tumour, small-cell lung cancer diagnosis
* Brainstem metastasis
* Leptomeningeal metastases
* Contraindication to MR imaging with contrast
* Pregnant or nursing women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with multiple (>= 4) brain metastases undergoing radiosurgery at the Winnipeg Centre for Gamma Knife Surgery.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2014-04; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Hopkins Verbal Learning Test - Revised (HVLT-R) | 4 months after radiosurgery

SECONDARY OUTCOMES:
Neurocognitive battery | 4 months after radiosurgery
  Other neurocognitive tests will include Trail making test A and B (TMT), Controlled Oral Word Association (COWAT), Test of Premorbid Functioning, Ruff Figural Fluency Test, Animal Naming, Brief Visuospatial Memory Test - Revised, WMS-III Digit Span, WMS-III Spatial Span, and the Symbol Digit Modalities Test.
Quality of Life | 4 months after radiosurgery
  * European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 15 Palliative (QLQ-C15-PAL)
  * Brain cancer specific quality of life questionnaire (QLQ-BN20)
Common Terminology Criteria for Adverse Events (CTCAE) v4.0 | 4 months after radiosurgery

OTHER OUTCOMES:
Time to in-field and distant radiographic progression | 1 year
Duration of functional independence (Barthel ADL index) | 1 year
Neurologic death rate | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Harvey Quon, MD, Principal Investigator — CancerCare Manitoba
Locations (1):
- Health Sciences Centre / CancerCare Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No